CLINICAL TRIAL: NCT04457141
Title: Study Electromyographic Activity of the Muscles of the Pelvic Floor Runners With Conventional Shoes and Minimalist.
Acronym: minimalwomen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 19/570-E_TFM
Record Dates: First submitted 2020-05-12; First posted 2020-07-07 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2021-11

CONDITIONS: Stress Urinary Incontinence
Keywords: Pelvic floor; Electromyography; Barefoot
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first:shod ,second:minimalist shoes (Other): The first group will race with conventional shoes and then minimalist shoes. The group run 5 minutes for warming and then 30 seconds at 6km/h, 30 seconds at 9 km/h and 30 seconds at 11km/h.
  They have a washout period of 10 minutes between both interventions.
  Interventions: Combination Product: Effect of pelvic floor for the use of minimalist shoes versus shod in woman.
- first:minimalist shoes ,second:shod (Other): The second group will race with minimalist shoes and then conventional shoes. The group run 5 minutes for warming and then 30 seconds at 6km/h, 30 seconds at 9km/h and 30 seconds at 11km/h.
  They have a washout period of 10 minutes between both interventions.
  Interventions: Combination Product: Effect of pelvic floor for the use of minimalist shoes versus shod in woman.

INTERVENTIONS:
Combination Product: Effect of pelvic floor for the use of minimalist shoes versus shod in woman. — Measure the activity of the pelvic floor and others muscles with EMG during treadmill running with different speeds and different shoes: minimalist and shod.

SUMMARY:
JUSTIFICATION:

Urinary incontinence is highly prevalent among women who play high impact sports such as running. that observed one of the possible reasons for this high prevalence is delayed activation of the pelvic floor in relation to the abdominal muscles.

The use of minimalist shoes during the race produces changes in muscle and joint biomechanics and efficiency in the race. However, to date no studies evaluating the influence of footwear in the musculature of the pelvic floor during the race.

OBJECTIVE: Describe and compare the electromyographic activity of the muscles of the pelvic floor and abdominal during the race with conventional shoes and minimalist.

DESIGN: cross-over study experimental, analytical and prospective. METHODOLOGY: conventional and minimalist: 50 healthy young women, 6- randomly distributed in two groups will be included to characterise the electromyographic activity of the pelvic floor muscles before and during running at 6-9-11 km/h with the two types of running shoes.

A baseline assessment will be performed to confirm that the women meet the inclusion and exclusion criteria. The ability to run a 10-minute treadmill at a speed of 6-9-11 km/h will be assessed, as well as the ability to adequately contract the pelvic floor muscles.

The group of 50 women will initially run randomly with conventional running shoes or with minimalist running shoes, and then, after a 10-minute washout period, will run with the other type of running shoe, i.e. if a participant in the first phase used conventional running shoes, she will run with a minimalist running shoe in the second phase.

The cadence of step, the range of movement of the femur and the EMG recording with electromyographic sensors of the pelvic floor musculature (using an intravaginal probe of the germproof brand), abdominal (internal and external oblique), spinal erectors and gluteus (using a surface sensor) in relation to the cycling gait will be collected and recorded with barographic sensors. The variables to be included in the electromyography for each muscle in relation to the gait cycle will be: onset of activation, duration, intensity and synergy with their corresponding standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 38 years.
* Nulliparous.
* Clinically healthy at the time of the study.
* Physically able for the requirement of the race on tape.
* Body Mass Index (BMI) 20-25 kg / m2
* Having signed the informed consent.

Exclusion Criteria:

* Pregnant women.
* urogynecological dysfunction.
* Lower limb surgeries performed in the last six months.
* Not be able to make voluntary contractions of the pelvic floor standardized according to the Modified Oxford Scale

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Electrical activation of the pelvic floor musculature, abdominal, gluteus maximus and lumbar erectors during the race in nulliparous women with sneakers traditional and minimalist | Basal, 0.5, 1.0, 1.5 minutes after the start of the test.
  PeriformTM vaginal probe Will collect the EMG activity of the muscles of the pelvic also register with superficial electrodes EMG abdominal, gluteus maximus and lumbar erectors. Records are made in a single session with washout periods in accordance with previous studies that have collected the activity of the EMG activity PF during treadmill running different speeds.

SECONDARY OUTCOMES:
Cadence and Range of motion in the sagittal plane of the femur during running at different speeds in nulliparous women with conventional and minimalist shoes. | Basal, 0.5, 1.0, 1.5 minutes after the start of the test.
  Collect of the spatial displacement of the lower limb by means of an accelerometer located in the EMG sensor during the treadmill race at different speeds
Maximum voluntary contraction (MVIC), minimum peak, maximum peak and total average of the muscles of the sp, abdominal (LE), gluteus maximus and erectors during running at different speeds in nulliparous women with conventional shoes and minimalist | Basal, 0.5, 1.0, 1.5 minutes after the start of the test.
  PeriformTM vaginal probe Will collect the EMG activity of the muscles of the pelvic also register with superficial electrodes EMG abdominal, gluteus maximus and lumbar erectors. Records are made in a single session with washout periods in accordance with previous studies that have collected the activity of the EMG activity PF during treadmill running different speeds.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Garcia, Principal Investigator — universidad complutense
Locations (1):
- Department of Radiology, Rehabilitation and Physiotherapy, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
All the researchers will participate in all the study phases.